CLINICAL TRIAL: NCT05757648
Title: Effect of Buffered Anesthetic on Physiological Reactions During Dental Injection in Young Children Under Deep Sedation: A Prospective, Single Visit, Randomized, Double-Blind Split Mouth Study
Brief Title: Buffered Local Anesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20191693
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Dental Pain
Keywords: Dental surgery; Deep sedation
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: Patients serve as their own control. One side of the mouth is buffered, one side is non-buffered
Masking Description: Participant and Care provider is blinded as to which side is buffered and which is non-buffered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Buffered Anesthetic Side/Non-buffered Anesthetic Side (Experimental): Patients will be randomized to one side of the mouth getting the buffered anesthetic and the other side of the mouth to the non-buffered anesthetic.
  Patients will be randomized to one side of the mouth getting the buffered anesthetic and the other side of the mouth to the non-buffered anesthetic.
  Interventions: Drug: Non-buffered Anesthetic; Drug: Buffered Anesthetic; Device: Onset

INTERVENTIONS:
Drug: Non-buffered Anesthetic — non-buffered LA, 2% lidocaine with epinephrine 1:100,000
Drug: Buffered Anesthetic — A cartridge of 2% lidocaine with epinephrine 1:100,000 alkalinized at 9:1 ratio with a resulting pH of 7.21 using 8.4% sodium bicarbonate solution per manufacturer.
Device: Onset — The test solution will be made by a mixing pen called "Onset"- This mixing pen Onset will deliver 0.18 mL of sodium bicarbonate solution into the anesthetic cartridge.

SUMMARY:
The purpose of this research study is to compare responses in children during dental injections of local anesthetic (used for numbing), while children are under deep sedation (breathing on their own, often with a loss of consciousness). Two types of local anesthetic will be used--one will be buffered (by adding a salt solution to make it less acidic), while the other will be plain, without anything added. Previous studies have shown that the addition of the buffer solution can improve comfort during a dental injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children or children with mild controlled systemic illness
* Treatment planned to receive restorative work on both sides of mouth (left vs right) under deep sedation, requiring local anesthetic administration

Exclusion Criteria:

* Children present with any illness or symptoms that can alter pain perception such as pain in head and neck area due to TMJ disorders, arthritis, autoimmune diseases
* Antibiotic premedication requirement
* History of taking medications (NSAIDs, narcotics, sedatives, and antianxiety or antidepressant medications) that may affect anesthetic assessment
* Has signs of dental pain, odontogenic abscess or facial cellulitis
* Allergy to local anesthetics or sulfites

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying An, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Dental Clinic of Rainbow Center for Women and Children, Cleveland, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Mouth Side
Groups:
- All Study Participants: Patients will be randomized to one side of the mouth getting the buffered anesthetic and the other side of the mouth to the non-buffered anesthetic.
  Non-buffered Anesthetic: non-buffered LA, 2% lidocaine with epinephrine 1:100,000
  Buffered Anesthetic: A cartridge of 2% lidocaine with epinephrine 1:100,000 alkalinized at 9:1 ratio with a resulting pH of 7.21 using 8.4% sodium bicarbonate solution per manufacturer.
  Onset: The test solution will be made by a mixing pen called "Onset"- This mixing pen Onset will deliver 0.18 mL of sodium bicarbonate solution into the anesthetic cartridge.
Period: Overall Study
Arm/Group | All Study Participants
Started | 20; 40 Mouth Side
Completed | 20; 40 Mouth Side
Not Completed | 0; 0 Mouth Side

BASELINE CHARACTERISTICS:
Groups:
- Buffered Anesthetic Side/Non-buffered Anesthetic Side: Patients will be randomized to one side of the mouth getting the buffered anesthetic and the other side of the mouth to the non-buffered anesthetic.
  Patients will be randomized to one side of the mouth getting the buffered anesthetic and the other side of the mouth to the non-buffered anesthetic.
  Non-buffered Anesthetic: non-buffered LA, 2% lidocaine with epinephrine 1:100,000
  Buffered Anesthetic: A cartridge of 2% lidocaine with epinephrine 1:100,000 alkalinized at 9:1 ratio with a resulting pH of 7.21 using 8.4% sodium bicarbonate solution per manufacturer.
  Onset: The test solution will be made by a mixing pen called "Onset"- This mixing pen Onset will deliver 0.18 mL of sodium bicarbonate solution into the anesthetic cartridge.
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Score as Measured by the Behavior Pain Scale
Description: The BPS score ranges from 2 to 8 points. The higher the score, the more potential pain an unconscious patient is experiencing during sedation procedures.
Time Frame: Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
score on a scale
  Buffered Anesthetic Side | 2.24 [2.06 to 2.42]
  Non-Buffered Anesthetic Side | 2.61 [2.42 to 2.79]
Statistical Analysis 1: Comparison: Buffered Anesthetic Side/Non-buffered Anesthetic Side; Test type: Superiority; p = 0.005, Mixed Models Analysis

2. Primary Outcome: Change in Heart Rate as Measured by as Measured by Medical Record
Time Frame: Baseline, Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
Beats per minute
  Baseline | 91 [86.6 to 95.4]
  10 minutes | 95 [90.6 to 99.4]
Statistical Analysis 1: Comparison: Buffered Anesthetic Side/Non-buffered Anesthetic Side; Test type: Superiority; p = 0.775, Mixed Models Analysis

3. Primary Outcome: Change in Diastolic Blood Pressure as Measured by Medical Record
Time Frame: Baseline, Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
mmHG
  Baseline | 52 [47.4 to 56.6]
  10 minutes | 53.2 [48.5 to 57.8]
Statistical Analysis 1: Comparison: Buffered Anesthetic Side/Non-buffered Anesthetic Side; Test type: Superiority; p = 0.682, Mixed Models Analysis

4. Primary Outcome: Change in Systolic Blood Pressure as Measured by Medical Record
Time Frame: Baseline, Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
mmHG
  Baseline | 91 [86.6 to 95.4]
  10 minutes | 95 [90.6 to 99.4]

5. Primary Outcome: Change in CO2 Level as Measured by Medical Record
Time Frame: Baseline, Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: mEq/L
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
mEq/L
  Baseline Buffered Side | 39.7 [37.2 to 42.1]
  Up to 10 mins Buffered Side | 40.3 [37.8 to 42.8]
  Baseline Non-Buffered Side | 40.9 [38.4 to 43.5]
  Up to 10 mins Non-Buffered Side | 40.2 [37.7 to 42.7]

6. Primary Outcome: Change in Oxygen Saturation Level as Measured by Medical Record
Time Frame: Baseline, Up to 10 minutes
Measure: Mean (95% Confidence Interval); unit: percentage of oxygen saturation
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
Number analyzed (Participants) | 20
percentage of oxygen saturation
  Baseline Buffered Side | 99.3 [98.6 to 100]
  Up to 10 mins Buffered Side | 99.0 [98.3 to 99.6]
  Baseline Non-Buffered Side | 99.4 [98.7 to 100]
  Up to 10 mins Non-Buffered Side | 99.2 [98.6 to 99.9]

ADVERSE EVENTS:
Time Frame: Monitored during post op only, up to 3 hours
Arm/Group | Buffered Anesthetic Side/Non-buffered Anesthetic Side
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05757648/Prot_SAP_000.pdf